CLINICAL TRIAL: NCT01357668
Title: An Observational Registry of Abatacept in Patients With Juvenile Idiopathic Arthritis
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-240
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with JIA who are treated with Abatacept: Patients with JIA who are treated with Abatacept according to physicians'/families' decisions

SUMMARY:
The purpose of this study is to examine the long-term safety of Abatacept for the treatment of juvenile idiopathic arthritis (JIA) with particular in interest in the occurrence of serious infections, autoimmune disorders, and malignancies.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria

* Diagnosis of JIA (any subtype)
* Age < 18 years at the time of enrollment unless currently or previously enrolled in an abatacept clinical trial and received abatacept
* Receiving Abatacept at the time of enrollment as per treating physician's decision or received abatacept in a clinical trial
* Parent or legally acceptable representative willing to participate in the study and sign the informed consent

Exclusion Criteria

* Pregnant or nursing female at the time of enrollment
* Prior malignancies if the patient has not been malignancy free for at least 5 years.
* Any serious acute or chronic medical condition other than JIA, including chronic infection, which would compromise the patient's ability to participate in the study
* Known poor compliance with clinic visits (based on physician judgment).

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric rheumatology clinics
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2013-01-30 (Actual); Primary Completion 2029-01-02 (Estimated); Study Completion 2029-01-02 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of serious infections | 10 years
Incidence rate of malignancies | 10 years
Incidence rate of autoimmune disorders | 10 years

SECONDARY OUTCOMES:
Number of serious adverse events | 10 years
Number of targeted infections (Epstein-Barr virus, cytomegalovirus, papilloma virus, herpes zoster, tuberculosis and opportunistic infections) | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (59):
- United States (3):
  - Local Institution - 0060, Little Rock, Arkansas
  - Local Institution - 0001, Princeton, New Jersey
  - Local Institution - 0059, Cincinnati, Ohio
- Austria (3):
  - Local Institution - 0025, Bregenz
  - Local Institution - 0002, Innsbruck
  - Local Institution - 0032, Vienna
- Brazil (4):
  - Local Institution - 0010, Botucatu, São Paulo
  - Local Institution - 0026, Campinas, São Paulo
  - Local Institution - 0028, São Paulo, São Paulo
  - Local Institution - 0027, Rio de Janeiro
- Canada (2):
  - Local Institution - 0029, Calgary, Alberta
  - Local Institution - 0011, Montreal, Quebec
- Denmark (2):
  - Local Institution - 0035, Aarhus, Central Jutland
  - Local Institution - 0012, Copenhagen
- France (3):
  - Local Institution - 0040, Clermont-Ferrand, Puy-de-Dôme
  - Local Institution - 0005, Paris
  - Local Institution - 0041, Toulouse
- Germany (5):
  - Local Institution - 0003, Bad Bramstedt
  - Local Institution - 0030, Berlin
  - Local Institution - 0034, Freiburg im Breisgau
  - Local Institution - 0031, Hamburg
  - Local Institution - 0033, Heidelberg
- Local Institution - 0016, Thessaloniki, Greece
- Local Institution - 0017, Budapest, Hungary
- Local Institution - 0014, Jerusalem, Israel
- Italy (6):
  - Local Institution - 0042, Florence
  - Local Institution - 0015, Genova
  - Local Institution - 0043, Naples
  - Local Institution - 0045, Napoli
  - Local Institution - 0044, Padua
  - Local Institution - 0046, Trento
- Local Institution - 0018, Riga, Latvia
- Local Institution - 0006, Guadalajara, Jalisco, Mexico
- Netherlands (2):
  - Local Institution - 0047, Rotterdam
  - Local Institution - 0019, Utrecht
- Norway (2):
  - Local Institution - 0048, Tromsø
  - Local Institution - 0049, Trondheim
- Peru (2):
  - Local Institution - 0007, Lima
  - Local Institution - 0050, Lima
- Local Institution - 0020, Lisbon, Portugal
- Puerto Rico (2):
  - Local Institution - 0023, Bayamón
  - Local Institution - 0056, Bayamón
- Local Institution - 0021, Cluj-Napoca, Romania
- Russia (4):
  - Local Institution - 0051, Moscow
  - Local Institution, Moscow
  - Local Institution - 0053, Saint Petersburg
  - Local Institution - 0052, Saratov
- Saudi Arabia (2):
  - Local Institution - 0055, Jeddah
  - Local Institution - 0024, Riyadh
- Local Institution - 0022, Piešťany, Slovakia
- South Africa (3):
  - Local Institution - 0009, Pretoria, Gauteng
  - Local Institution - 0057, Panorama, Cape Town, Western Cape
  - Local Institution - 0058, Pretoria
- Spain (5):
  - Local Institution - 0036, Sant Joan Despí, Barcelona
  - Local Institution - 0004, Barcelona
  - Local Institution - 0038, Madrid
  - Local Institution - 0037, Murcia
  - Local Institution - 0039, Valencia
- Local Institution - 0013, Bristol, United Kingdom

REFERENCES:
- [Derived] Lovell DJ, Tzaribachev N, Henrickson M, Simonini G, Griffin TA, Alexeeva E, Bohnsack JF, Zeft A, Horneff G, Vehe RK, Stanevica V, Tarvin S, Trachana M, Del Rio AQ, Huber AM, Kietz D, Orban I, Dare J, Foeldvari I, Quartier P, Dominique A, Simon TA, Martini A, Brunner HI, Ruperto N; for PRINTO and the Pediatric Rheumatology Collaborative Study Group (PRCSG) section sign. Safety and effectiveness of abatacept in juvenile idiopathic arthritis: results from the PRINTO/PRCSG registry. Rheumatology (Oxford). 2024 Sep 1;63(SI2):SI195-SI206. doi: 10.1093/rheumatology/keae025. PMID 38243722
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html